CLINICAL TRIAL: NCT04989543
Title: Study of the Composition and Bacterial Diversity of the Vaginal Microbiota in Healthy Versus Pathological Conditions (Bacterial Vaginosis) Using a Targeted Metagenomic Approach (RNA 16s)(CEBAM)
Brief Title: Study of the Composition and Bacterial Diversity of the Vaginal Microbiota in Healthy Versus Pathological Conditions (Bacterial Vaginosis) Using a Targeted Metagenomic Approach (RNA 16s)
Acronym: CEBAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Larena SAS (Industry)
Collaborators: CEN Biotech (Industry); Luxia Scientific (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: C1664
Record Dates: First submitted 2021-03-10; First posted 2021-08-04 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-04

CONDITIONS: Vaginosis, Bacterial
Keywords: Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- healthy population (Other): Interventions: vaginal swabs:
  * Nugent scores,
  * cytobacteriological examination (in particular to determine the "Clue Cells")
  * evaluation of the vaginal microbiota.
  On receipt of the Nugent score results, the doctor will confirm whether or not the patient is included in one of the two arms under study:
  * healthy" population
  * pathological" population with bacterial vaginosis
  Interventions: Diagnostic Test: vaginal swabs
- pathological population (Other): Interventions: vaginal swabs:
  * Nugent scores,
  * cytobacteriological examination (in particular to determine the "Clue Cells")
  * evaluation of the vaginal microbiota.
  On receipt of the Nugent score results, the doctor will confirm whether or not the patient is included in one of the two arms under study:
  * healthy" population
  * pathological" population with bacterial vaginosis
  Interventions: Diagnostic Test: vaginal swabs

INTERVENTIONS:
Diagnostic Test: vaginal swabs — Nugent score: Vaginal swabbing with the dry swab, make two smears on slides.
  Cytobacteriological examination: swabbing at the exo-endocrine junction using the swab
  Evaluation of the vaginal microbiota: swabbing at the exo-endocrine junction using the swab

SUMMARY:
It aims to determine and compare the degree of vaginal bacterial alpha diversity in the absence (healthy population) or presence of bacterial vaginosis (pathological population).

ELIGIBILITY:
Inclusion Criteria:

* Woman aged between ≥ 18 and ≤ 45 years old,
* In good general health (outside the gynaecological sphere), i.e. no chronic pathology and not taking medication at the time of inclusion and/or long-term,
* Woman with a healthy or pathological vaginal flora according to Amsel's clinical diagnosis and Nugent's score :

Population with bacterial vaginosis (verification of at least the following 3 criteria + Nugent score):

* Vaginal pH > 4.5
* greyish, homogenous vaginal secretions adhering to the vaginal wall
* characteristic vaginal odour of "rotten fish" after contact of the vaginal discharge with a few drops of 10% potash ("sniff test")
* Presence of "Clue Cells" in the microscopic examination of fresh vaginal secretions. Clue cells are cells of the ectocervix lined with gram-negative bacilli.

  * Nugent Score ≥ 7

Healthy population (Verification of at least 3 following criteria + Nugent score) :

* Absence of vaginal pH > 4.5
* No greyish, homogenous vaginal secretions adhering to the vaginal wall
* No characteristic vaginal odour of "rotten fish" after contact of the vaginal discharge with a few drops of 10% potash ("sniff test").
* Absence of "Clue Cells" on microscopic examination of fresh vaginal secretions. Clue cells" are cells of the ectocervix lined with gram-negative bacilli.

  * Nugent Score ≤3

    * Able and willing to participate in the research by complying with the procedures of the protocol, especially regarding vaginal sampling,
    * Having given its free, informed and written consent.

Exclusion Criteria:

* Patient during menstruation,
* Patient who has had vaginal sex within 48 hours,
* Patient with irregular menstrual cycles,
* Patient undergoing preventive or curative treatment for vaginal infections,
* Patients suffering from other diseases of the vagina (herpes, chlamydia, syphillis),
* Patients undergoing antibiotic or antifungal treatments or taken less than 3 months ago,
* Patient under probiotic or prebiotic complementation or taken less than a month ago,
* Patient with systemic or immunodeficient disease,
* Patient with an alcohol consumption of more than 2 glasses per day,
* Pregnant or breastfeeding woman, or woman planning to become pregnant within the next 8 weeks, or woman in the post-partum period,
* Patient unable to understand information related to the study (mental or linguistic disability),
* Patient participating or having participated within the previous 3 months in another clinical trial, or in a period of exclusion from a clinical trial,
* Patient not affiliated to a social security scheme.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2021-11-03 (Actual)

PRIMARY OUTCOMES:
Determine and compare the degree of vaginal bacterial alpha diversity in the absence (healthy population) or presence of bacterial vaginosis (pathological population). | Day 0
  The degree of vaginal bacterial alpha diversity in healthy and pathological conditions (bacterial vaginosis) will be evaluated by the Shannon index. It will be determined by the identification of the bacterial species (16s RNA analysis) present on a vaginal swab taken during the selection visit.

SECONDARY OUTCOMES:
Determine and compare in healthy versus pathological conditions (bacterial vaginosis) : - vaginal specific richness in enterotypes, - The diversity of vaginal bacterial species by other indices, - The overall composition of the vaginal microbiota. | Day 0
  * Enterotypic richness will be assessed by 16 S analyses on the vaginal swab taken during the selection visit.
  * The α-diversity will be calculated using other indices.
  * The overall composition of the vaginal microbiota will be assessed from a taxonomic point of view on the vaginal swab taken during the selection visit by calculating the percentage (relative quantification).

OTHER OUTCOMES:
- Identify threshold values of bacterial diversity beyond which a bacterial vaginosis would be established; - Validate these thresholds by comparison with the Nugent score and the Amsel diagnosis. | Day 0
  The possible thresholds of bacterial diversity above which bacterial vaginosis is observed will be validated by comparison with the Nugent score made during the screening visit and the Amsel diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Samira AIT ABDELLAH, Study Director — Larena SAS
Locations (1):
- Institut FOURNIER, Paris, France

IPD SHARING:
Plan to Share IPD: No